CLINICAL TRIAL: NCT03657394
Title: A Cluster Randomized Clinical Trial of Umbilical Cord Milking Versus Early Cord Clamping on Short and Long-term Outcomes in Neonates Who Are Non-Vigorous at Birth
Brief Title: Comparative Outcomes Related to Delivery-room Cord Milking In Low-resourced Kountries
Acronym: CORDMILK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Sharp HealthCare (Other); Thomas Jefferson University (Other); University of San Diego (Other); St. Louis University (Other); Jawaharlal Nehru Medical College (Other); Daga Memorial Maternity and Children's Hospital, Nagpur, India (Unknown); Mahatma Gandhi Institue of Medical Sciences, Wardha, India (Unknown); Karnataka Institue of Medical Sciences, Hubbali, India (Unknown); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); All India Institute of Medical Sciences (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Indira Gandhi Government Medical College & Hospital, Nagpur, India (Unknown); Pimpri Chinchwad Municipal Corporation's Post-Graduate Institute, Yashwantrao Chavan Memorial Hospital, Pune, India (Unknown); Government Medical College, Nagpur (Industry)
Responsible Party: Principal Investigator, Zubair Aghai, Professor Of Pediatrics, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CORDMILK; R01HD102967 (NIH)
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Birth Asphyxia
Keywords: Placental transfusion
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Crossover
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): The delivering practitioner will place the newborn below the level of the incision (at the edge of the table) at C/S and a second team member will milk the cord four times. For vaginal delivery, the delivering obstetrician, midwife or perinatal provider will hold the infant against their body or place the infant on the mother's abdomen and the cord will be milked either four times by the obstetrical provider or by a second team member. For the cord milking procedure, the obstetrical provider will milk 20-30 centimeters length of the umbilical cord over two seconds, repeating three additional times as described previously. This time is not significantly different from the time for ECC.
  Interventions: Other: Umbilical cord milking
- Early Cord Clamping (No Intervention): Umbilical cord will be clamped immediately after birth (within 60 seconds)

INTERVENTIONS:
Other: Umbilical cord milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 1--15 seconds.
  Arms: Umbilical Cord Milking

SUMMARY:
The investigators will conduct a study on non-vigorous infants at birth to determine if umbilical cord milking (UCM) results in lower rate of moderate to severe hypoxic ischemic encephalopathy (HIE) or death than early clamping and for infants who are non-vigorous at birth and need immediate resuscitation.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a brain injury caused by inadequate blood flow and oxygen delivery to the neonatal brain. Almost all infants with severe HIE and 30-50% infants with moderate HIE either die or develop significant developmental delay, cerebral palsy or other disabilities.The incidence of HIE is 1-3 per 1,000 term births in developed countries and 15-20 times higher in developing countries (Worldwide, 0.5 to 1 million infants develop HIE each year). Therapeutic hypothermia is the only proven therapy for infants with HIE. Even after receiving therapeutic hypothermia, one-half of all infants with moderate and severe HIE die or develop neurological and functional impairment. Therapeutic hypothermia is not widely available and ineffective in developing nations.There is an urgent need for a new therapy for neonates with HIE, which can complement hypothermia and be readily available in developing nations. Stem cell transplantation is a potential therapy for infants with HIE. Umbilical cord blood is a rich source of stem cells. Umbilical cord milking (UCM) may have similar effect as autologous umbilical cord blood cell transplantation.

Preliminary evidence suggests a placental transfusion in term infants may be a neuroprotective mechanism that can also facilitate cardiovascular transition for neonates depressed at birth and result in decreased mortality and improved neurodevelopmental outcomes. Infants with HIE, due to varied complications during the birth process, have poor perfusion due to fetal blood volume loss to the placenta. However, the most common method of providing placental blood, delayed cord clamping (DCC) cannot be performed since infants with HIE are non-vigorous and providers often need to perform resuscitation immediately after birth. The World Health Organization and the American College of Obstetrics and Gynecology (ACOG) also does not recommended DCC in neonates who are non-vigorous (limp, pale, and not breathing) at birth and require immediate resuscitation. Umbilical cord milking (UCM) or gently squeezing cord blood toward the baby, is an alternative to DCC, which can achieve significant placental transfusion without delaying resuscitation. Further, UCM can be completed as quickly as immediate cord clamping (ICC) and UCM requires minimal training and no additional staff.

The investigators hypothesized that UCM will reduce the number of infants developing moderate to severe HIE or death in neonates who are non-vigorous at birth compared to early cord clamping (ECC). This will be a cluster crossover randomized controlled trial. Each hospital will be randomly assigned to use either ECC or UCM for any infant who is non-vigorous at birth and needing resuscitation over a period of 6 months. Then the site will change to the other method for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-vigorous neonates born between 35-42 weeks

Exclusion Criteria:

* Congenital malformation of CNS.
* Chromosomal abnormalities.
* Major congenital malformations.
* Abruption/cutting through the placenta at delivery.
* Umbilical cord knots or inadequate cord length.
* Mono-chorionic twins or twins with no information on amnion/chorion.
* Multiple gestation >2 .

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3442 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Moderate to severe HIE or death | From date of birth until the date of discharge from the hospital or date of death from any cause, whichever come first, asessed up to 10 weeks.
  Number of infants with moderate to severe HIE or death

SECONDARY OUTCOMES:
MRI of the brain | 4 days to 2 weeks
  Number of infants with moderate to severe HIE who have abnormal brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Zubair H Aghai, MD, Principal Investigator — Nemours Children's Clinic; Anup Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns; Sangappa Dhaded, MD, Principal Investigator — KLE Academy of Higher Education and Research
Locations (9):
- India (9):
  - KLE Academy of Higher Education and Research (Deemed-to-be-University) Jawaharlal Nehru Medical College, Belagavi, Karnataka
  - Indira Gandhi Government Medical College & Hospital, Nagpur, Maharashtra
  - Pimpri Chinchwad Municipal Corporation's Post-Graduate Institute, Yashwantrao Chavan Memorial Hospital, Pune, Maharashtra
  - Government Medical College, Chandrapur, MS
  - Daga Memorial Woman and Children Hospital, Nagpur, MS
  - Government Medical College and Hospital, Nagpur, MS
  - All India Institute of Medical Science, Nagpur, MS
  - Mahatma Gandhi Institute of Medical Sciences/ Kasturba Hospital, Wardha, MS
  - Sawai Man Singh (SMS) Medical College, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yogeshkumar S, Vernekar SS, Dhaded SM, Talekar K, Leiby BE, Hartman R, Vaucher Y, Chouthai N, Girish M, Jain M, Jain S, Parvekar S, Jain V, Patankar A, Suryawanshi M, Tiwari M, Waikar M, Nashine N, Ambike D, Asalkar M, Kulkarni R, Haribhaktha S, Narkhede H, Chaudhari S, Kamble M, Shrirame D, Falke B, Mehta S, Verma A, Gothwal S, Goudar SS, Derman R, Katheria A, Aghai ZH. CORDMILK: Umbilical Cord Milking versus Early Cord Clamping on short-and long-term outcomes in neonates who are non-vigorous at birth-study protocol of a multi-center, cluster-randomized, crossover-controlled trial. Trials. 2025 Nov 17;26(1):509. doi: 10.1186/s13063-025-09197-8. PMID 41250198